CLINICAL TRIAL: NCT03425344
Title: Discriminative Validity of Real-time Sonoelastography of the Supraspinatus Tendon: Comparison of Findings Between Patients With Supraspinatus Tendinopathy and Healthy Volunteers
Brief Title: Discriminative Validity of Strain Elastography of the Supraspinatus Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Brage (Other)
Collaborators: Odense University Hospital (Other); Sygehus Lillebaelt (Other); Gigtforeningen (Other); Region of Southern Denmark (Other); Radiograf Rådet (Unknown)
Responsible Party: Sponsor-Investigator, Karen Brage, Ph.D-student, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SEL_Supraspinatus_cross
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Elasticity Imaging Techniques; Tendinopathy; Rotator Cuff Tendinitis; Musculoskeletal Disease
MeSH Terms: conditions — Tendinopathy; Rotator Cuff Injuries; Musculoskeletal Diseases | interventions — Diagnosis

STUDY DESIGN:
Intervention Model Description: A case-control study without intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Other): All participants will be exposed to shoulder- MRI, ultrasound and sonoelastography.
  Interventions: Diagnostic Test: Diagnostic

INTERVENTIONS:
Diagnostic Test: Diagnostic — No traditionally intervention will be given but participants will be exposed to shoulder- MRI, ultrasound and sonoelastography..

SUMMARY:
This study aims at testing the discriminative validity of strain elastography in the normal and abnormal/pathological Supraspinatus tendon due to tendinopathy

DETAILED DESCRIPTION:
The case-control trial will include 96 participants. 48 of them diagnosed with supraspinatus tendinopathy by MRI and 48 healthy subjects.

In this study the investigators will compare the outcome of tissue elasticity measured by sonoelastography, with MRI and conventional ultrasound.

Patients will be recruited through different radiology department and healthy volunteers will be recruited primarily through advertising in local newspapers and social media.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30
* Symptomatic: Positive on 3/5 clinical tests (full can, empty can, resisted external rotation, neers, hawkins.
* Asymptomatic: No shoulder pain in the last year, negative on 5/5 clinical tests (full can, empty can, resisted external rotation, neers, hawkins).

Exclusion Criteria:

* Shoulder-fracture, operation and luxation, known-neuromuscular disease, rheumatoid arthritis, cancer, fibromyalgia, spondyloarthropathy and psychiatric disorders, pregnancy and inability to read and understand Danish. Biceps rupture, labrum lesions, supraspinatus tears (> 1/3 of the vertical tendon height) and calcifications (> 2 mm in length) (MRI).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Tendon quality (SEL) | Baseline
  Sonoelastography - strain elasticity

SECONDARY OUTCOMES:
Pain on a VAS scale | Baseline
  Change from baseline in Visual Analogue Scale (VAS). Ranging from 0 to 10; 0 being no pain and 10 being severe pain.
Quality of life on the E!-5D-3L questionnaire | Baseline
  Change in Euro Qol 5D index (EQ-5D-3L). The system consists of a descriptive system and a visual analogue scale (EQ VAS). The descriptive system contains 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 3 levels; no problems, some problems and extreme problems. The EQ-VAS range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Disability | Baseline
  Change in Disability of the Arm, Shoulder and Hand questionnaire (DASH). Each item is rated with a score from 1 (least disability) to 5 (most disability). All scores are added together, producing a raw score, which is then transformed into a score of 100 maximum. A higher score indicates greater disability.
Tendon quality (MRI) | Baseline
  Magnetic Resonance
Tendon quality (US) | Baseline
  Conventional ultrasound

OTHER OUTCOMES:
Demographic | Baseline
  Gender, age, bmi, education (level), duration of symptoms, symptom history

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Juul-Kristensen, Assoc. Prof, Study Director — Department of Sport Science and Biomechanics
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No